CLINICAL TRIAL: NCT02895815
Title: A Phase 2, Multicenter, Randomized Study Evaluating the Efficacy and Safety of Subretinal Administration of CNTO 2476 in Subjects With Visual Acuity Impairment Associated With Geographic Atrophy (GA) Secondary to Age Related Macular Degeneration (AMD)
Brief Title: Efficacy and Safety Study of CNTO 2476 in Participants With Visual Acuity Impairment Associated With Geographic Atrophy (GA) Secondary to Age Related Macular Degeneration (AMD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company business decision
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR108188; CNTO2476MDG2003 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-08-19; First posted 2016-09-12 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Visual Acuity; Geographic Atrophy; Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CNTO 2476 (6.0 * 10^4 cells) (Experimental): Participants will receive a single subretinal administration of CNTO 2476 (6.0 * 10^4 cells) in 50 microliter (mcL) given by subretinal delivery system.
  Interventions: Combination Product: CNTO 2476 (6.0 * 10^4 cells)
- CNTO 2476 (3.0 * 10^5 cells) (Experimental): Participants will receive a single subretinal administration of CNTO 2476 (3.0 * 10^5 cells) in 50 mcL given by subretinal delivery system.
  Interventions: Combination Product: CNTO 2476 (3.0 * 10^5 cells)
- Control Group (No Intervention): Participants will undergo observations without surgery.

INTERVENTIONS:
Combination Product: CNTO 2476 (6.0 * 10^4 cells) — Participants will receive a single subretinal administration of CNTO 2476 (6.0 * 10^4 cells) in 50 mcL given by subretinal delivery system (subretinal access kit [SRAK-02 kit] and third arm accessory).
  Arms: CNTO 2476 (6.0 * 10^4 cells)
Combination Product: CNTO 2476 (3.0 * 10^5 cells) — Participants will receive a single subretinal administration of CNTO 2476 (3.0 * 10^5 cells) in 50 mcL given by subretinal delivery system (SRAK-02 kit and third arm accessory).
  Arms: CNTO 2476 (3.0 * 10^5 cells)

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of CNTO 2476 cells administered into the subretinal space by the suprachoroidal surgical approach and the subretinal access kit (SRAK-02) in participants with visual acuity impairment associated with Geographic Atrophy (GA) secondary to Age Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
This is a Phase 2 study to evaluate the efficacy and safety of a single subretinal administration of CNTO 2476 compared with the untreated control group, as well as to assess the safety and usability profile of the procedure and the device for cell therapy delivery in participants with visual acuity impairment associated with Geographic Atrophy (GA) secondary to Age Related Macular Degeneration (AMD). The duration of participation in the study for each participant is approximately 3 years. Efficacy will be evaluated at 6 month, 12 months and every 6 month thereafter. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a suitable candidate for ophthalmologic surgery, is willing and able to comply with the surgical procedure, scheduled visits, treatment plan, laboratory tests and other study procedures. Participant has met criteria of the surgery center anti coagulation protocol, if applicable
* Confirmed diagnosis of geographic atrophy (GA) secondary to age-related macular degeneration (AMD) confirmed within 28 days prior to initial randomization by the central reading center using fundus photographs and including the following; a) The study eyes must have at least 1 GA lesion that involves the fovea, and a Macular Photocoagulation Study (MPS) disc areas (DA) of >= 1 and <= 7 (1 Macular Photocoagulation Study Disc Area (MPS DA equivalent to 2.54 millimeter (mm)^2 on the retina) determined by screening images of fundus autofluorescence photographs as calculated by the reading center. If GA is multifocal, at least 1 lesion must be >= 0.5 DA, b) GA must be able to be photographed in its entirety and may be contiguous with peripapillary atrophy, c) Retinal photographs, fundus autofluorescence images, and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice, can be obtained d) The imaging center must be able to delineate and confirm peripapillary atrophy with fundus photography and fundus autofluorescence, e) Images must include the central field 1, 2, and 3 field images as defined by the University of Wisconsin standards as well as a supero temporal image to capture the subretinal injection area if possible
* Female participants must be postmenopausal with last menses 12 months prior, or longer without medical reasons (example, treatment with a drug), or a measured follicle stimulating hormone >= 26 milli-international units per milliliter (mIU/mL)
* Study eyes will have a best corrected visual acuity (BCVA) of 20/80 to 20/800 (Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR value 0.6-1.6). BCVA in the study eye must be worse than the BCVA in the fellow eye at screening
* Male participants must be sterile or willing to use 2 approved methods of contraception from first day postoperatively to 3 months postoperatively

Exclusion Criteria:

* Participant has a history of neovascular ("wet") AMD in the study eye, including any evidence of retinal pigment epithelium rips or evidence of subretinal or choroidal neovascularization. History or evidence of neovascular AMD in the fellow eye is allowed, if antivascular endothelial growth factor (VEGF) therapy has not been required for at least 8 weeks prior to screening
* A diagnosis of glaucoma with an intraocular pressure (IOP) >= 25 millimeter of mercury (mm Hg) while being treated with an ocular hypotensive drug. Treatment should be no more than 1 drug preparation/combination, which can contain 1 or 2 ocular hypotensive active ingredients; participants receiving more than 2 ocular hypotensive active ingredients are excluded
* Nuclear sclerotic cataract, cortical spoking, posterior subcapsular cataract above Grade 2 per Age Related Eye Disease Study (AREDS) scale or any other ophthalmologic condition that reduces the clarity of the media that, in the opinion of the investigator or reading center, interferes with ophthalmologic examination (example, corneal abnormalities, inadequate pupillary dilation)
* Myopia >-8 diopters and participants with >4 diopters of astigmatism, and >+10 diopters of hyperopia
* Previous vitrectomy, retinal detachment repair, submacular surgery, other surgical interventions targeting AMD, scleral buckling or glaucoma filtration surgery or any other extraocular or orbital procedure in the study eye that, in the opinion of the surgeon, would hamper the suprachoroidal cannulation procedure in the study eye

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-09 (Estimated); Primary Completion 2021-02-20 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Showing Improvement From Baseline of Greater Than or Equal to (>=) 15 Letters in Best Corrected Visual Acuity (BCVA) at Month 6 | Month 6
  The BCVA testing performed after refraction and under standardized photopic lighting conditions and distance using an Early Treatment Diabetic Retinopathy Study (ETDRS) log of the minimum angle of resolution (logMAR chart). The ETDRS chart at 4 meters is considered the 'gold standard' for visual acuity testing in clinical research for its physical and statistical properties.

SECONDARY OUTCOMES:
Percentage of Participants Showing Improvement >=15 BCVA Letters From Baseline at 12 Month | Baseline and Month 12
  Percentage of Participants Showing Improvement >=15 BCVA Letters From Baseline at 12 Month
Percentage of Participants Losing >=15 Best Corrected Visual Acuity (BCVA) Letters From Baseline at 6 and 12 Months | Baseline, Month 6 and 12
  Percentage of Participants Losing >=15 Best Corrected Visual Acuity (BCVA) Letters From Baseline at 6 and 12 Months
Change in Mean Number of BCVA Letters From Baseline at 6 and 12 Months | Baseline, Month 6 and 12
  Change in Mean Number of BCVA Letters From Baseline at 6 and 12 Months
Change in Growth Rate of Geographic Atrophy (GA) Lesion Documented at Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  The area of GA is determined based primarily on fundus autofluorescence (FAF) as well as fluorescein angiography and fundus photography.
Mean Change in Reading Acuity (RA) From baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Minnesota reading test will be used to determine RA measured in log of the minimum angle of resolution (logMAR).
Mean Change in Maximum Reading Speed (MRS) From Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Minnesota reading test will be used to determine maximum reading speed (MRS, [measured in characters per minute]).
Mean Change in Critical Print Size (CPS) From Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Minnesota reading test will be used to determine CPS measured in log of the minimum angle of resolution (logMAR).
Mean Change in Low Luminance Best Corrected Visual Acuity (LL BCVA) Letters From Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Low Luminance BCVA indicates the best possible vision that an eye can achieve with the use of trial frames/lenses following refraction under low luminance conditions.
Percentage of Participants With Gain of >= 15 Letters in LL BCVA From Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Percentage of Participants With Gain of >= 15 Letters in LL BCVA From Baseline to 6 and 12 Months
Mean Change in Contrast Sensitivity From Baseline to 6 and 12 Months | Baseline, Month 6 and 12
  Mean Change in Contrast Sensitivity From Baseline to 6 and 12 Months
Number of Participants With Significant Changes in Retinal Morphology | Baseline, Month 6 and 12
  Number of Participants With Significant Changes in Retinal Morphology
Percentage of Participants who Convert to Neovascular Age-Related Macular Degeneration (AMD) in the Study Eye and in the Fellow Eye | Baseline, Month 6 and 12
  Percentage of Participants who Convert to Neovascular Age-Related Macular Degeneration (AMD) in the Study Eye and in the Fellow Eye
Percentage of Participants who Achieved Technical Success in the Active Drug Group | 6 Months
  Percentage of participants who achieved technical success in the active drug group will be evaluated and the criteria that must be met to achieve technical success are :1) The device was accessible to the suprachoroidal space, 2) Micro needle reached to the subretinal space, 3) When study drug injected into the subretinal space a) No retinal perforation was directly visualized by the surgeon following the formation of the bleb in the subretinal space after injecting the balanced salt solution (BSS) Plus, b) When 50 microliter (mcL) of study drug was administered subretinally, the creation of an enlarged bleb in the subretinal space is visualized by the surgeon, 4) Micro needle and the device were removed.
Percentage of Participants who Achieved Procedural Success in the Active Drug Group | Month 6 and 12
  Percentage of participants who achieved procedural success in the active drug group will be evaluated and the criteria that must be met to achieve procedural success : 1) Achievement of technical success, 2) Endophthalmitis, significant choroidal hemorrhage, leakage of cells or other need for vitrectomy, retinal detachment, and failure to deliver cells did not occur, 3) No device malfunction.
Number of Participants with Ocular Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Long term Follow up (Month 36)
  Study treatment, device and surgical procedure-related ocular AEs and SAEs will be reported.
Mean Change From Baseline at 6 and 12 Months in Participants Reported Health-Related Quality of Life as Assessed by Short Form (36) Health Survey | Baseline, Month 6 and 12
  SF-36 is scored to produce 8 subscales (Physical Functioning, Role Limitations-Physical, Bodily Pain, General Health Perceptions, Vitality, Social Functioning, Role Limitations- Emotional, and Mental Health) and 2 summary scores (Physical Component Summary and Mental Component Summary).
Mean Change From Baseline at 6 and 12 Months in Participants Reported Health Related Quality of Life as Assessed by Functional Reading Index Questionnaire (FRI) | Baseline, Month 6 and 12
  The FRI is an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD participants. Item scores reflect decreasing levels of functional reading independence. The FRI Index yields continuous mean scores (range 1 to 4), and ordinal-level scores from Level 1 = "Unable to do" to Level 4 = "Totally independent." For each FRI Index reading activity performed in the past 7 days, participants are asked about the extent to which they required vision aids, adjustments in the activity, or help from another person.
Incidence of Anti-CNTO 2476 Antibodies | Baseline, Day 7 and 15, Month 2, 3 and 6
  Number of participants who develop antibodies.
Mean Change From Baseline at 6 and 12 Months in Participants Reported Health-Related Quality of Life as Assessed by National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) Score | Baseline, Month 6 and 12
  The 2000 version of the NEI-VFQ-25, which must be interviewer-administered, includes 25 items and is scored to produce 11 subscales and a general health item. The 11 subscales include General Vision (1 item), Ocular Pain (2 items), Near Activities (3 items), Distance Activities (3 items), Social Functioning (2 items), Mental Health (2 items), Role Difficulties (2 items), Dependency (3 items), Driving (3 items), Color Vision (1 item), and Peripheral Vision (1 item). Response to each question converted to 0-100 score. Each subscale, total score equal to (=) average of items contributing to score. For each subscale and total score, score range: 0 to 100, higher score equal to less symptoms/better visual functioning.
Mean Change From Baseline at 6 and 12 Months in Participants Reported Health-Related Quality of Life as Assessed by Near Vision Subscale Score | Baseline, Month 6 and 12
  A 3-item Near Vision subscale score of National Eye Institute will evaluate quality of life. Response to each question converted to 0-100 score. Each subscale, total score equal to average of items contributing to score. For each subscale and total score, score range: 0 to 100, higher score equal to less symptoms/better visual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.